CLINICAL TRIAL: NCT05896969
Title: Phase 1, Single Multiple Dose Escalation Study in a Randomized, Double-blind, Placebo Controlled Design to Investigate Safety, Tolerability, PK and PD of SC Administered SNK-396 in Subjects With Elevated Low-Density Lipoprotein Cholesterol
Brief Title: Dose Escalation of SNK-396 in Participants With Elevated Low-Density Lipoprotein Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: SynerK Pharmatech (Suzhou) Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNK-396-101
Record Dates: First submitted 2023-03-14; First posted 2023-06-09 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Elevated Low-Density Lipoprotein Cholesterol

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, multi-center, randomized, double-blind, placebo-controlled single and multiple dose escalation study with SC doses of SNK-396 in participants with elevated LDL-C. The study will be divided into two parts:
  * SAD cohorts;
  * MAD cohorts. The two parts will be completed sequentially. The MAD part may be initiated when safety, tolerability, and PK data are known and deemed acceptable for single doses of at least the 5 planned dose levels of the SAD cohorts.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD Cohort (Experimental): SAD Cohort 1 - 8 : Subjects in each cohort will be randomised will receive a single SC dose of SNK-396 within the dose range of 25 to 800 mg, or matching placebo.
  Interventions: Drug: SNK-396 - SAD cohort
- MAD cohort (Experimental): MAD Cohort 1 - 8 : Subjects in each cohort will be randomized will receive the active SNK-396 with dose range of SNK-396 anticipated to be from 25 to 800 mg or matching placebo
  Interventions: Drug: SNK-396 - MAD Cohort

INTERVENTIONS:
Drug: SNK-396 - SAD cohort — A single dose of SNK-396 within the dose range of 25 to 800 mg, or matching placebo.
  Arms: SAD Cohort
Drug: SNK-396 - MAD Cohort — Multiple doses of SNK-396 within the dose range of from 25 to 800 mg, or matching placebo.
  Arms: MAD cohort

SUMMARY:
This is a Phase 1, multi-center, randomized, double-blinded, placebo-controlled single and multiple dose escalation study with SC doses of SNK-396 in participants with elevated LDL-C. The study will be divided into two parts:

* SAD cohorts
* MAD cohorts

DETAILED DESCRIPTION:
The SAD part will consist of up to 8 cohorts of eligible participants with elevated LDL-C as defined as serum LDL levels between 2.6 - 4.9 mmol/L (inclusive)

The MAD part will consist of up to 8 cohorts of eligible participants with elevated LDL-C as defined as serum LDL levels between 2.6 - 4.9 mmol/L (inclusive)

ELIGIBILITY:
Inclusion Criteria -

1. Male or female, ≥18 and ≤65 years of age, with BMI ≥18.5 and ≤35.0 kg/m2.
2. Participants must be either non smoking (no use of tobacco or nicotine products within 3 months prior to screening) or social smoker as defined by smoking no more than 5 cigarettes (or nicotine equivalent) a week and no smoking during screening period or on study.
3. Participants must be with elevated LDL-C defined as serum LDL levels between 2.6 - 4.9 mmol/L (inclusive) at screening.
4. Healthy (except for the LDL-C status) participants.
5. Participants must have fasting triglyceride level <4.52 mmol/L (<400mg/dL) at screening.
6. Sexually active females of childbearing potential and non-sterile males must be willing to use an acceptable contraceptive method throughout the study as detailed in section 8.1.
7. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria -

1. Any clinically significant abnormal finding at physical examination in the opinion of the investigator.
2. Subjects with a history or presence of cardiovascular disease (including cerebrovascular accident (stroke or TIA) or disease, uncontrolled hypertension, familial hypercholesterolaemia, obstructive sleep apnoea, and peripheral artery), a diagnosis of diabetes mellitus given potential for hyperglycaemia defined as HbA1c greater or equal to 6.5%, or a non-alcoholic fatty liver disease.
3. Received Leqvio (inclisiran) treatment in less than 6 months ago.
4. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | SAD - Up to Day 57 (end of study visit)
  Number of Subjects with Treatment Emergent Adverse Events
Treatment emergent adverse events | MAD - Up to Day 85 (end of study visit)
  Number of Subjects with Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  Cmax will be assessd
Pharmacokinetic Assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  tmax will be assessd
Pharmacokinetic Assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  AUC will be assessd
Pharmacokinetic Assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  T 1/2 will be assessd
Pharmacodynamic (PD) effect assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  LDL-C serum concentration will be assessed.
Pharmacodynamic (PD) effect assessment | Upto Day 57 for SAD , Upto Day 85 for MAD
  PCSK9 plasma levels concentration will be assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Nucleus Network Pty Ltd, Herston, Queensland
  - Cmax Clinical Research, Adelaide, South Australia
  - Nucleus Network Pty Ltd, Melbourne, Victoria